CLINICAL TRIAL: NCT03972267
Title: Influence of Enamel Matrix Derivative (Emdogain®) on Palate Wound Healing. Randomized Clinical Trial
Brief Title: Influence of Enamel Matrix Derivative (Emdogain®) on Palate Wound Healing.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, assistant professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF10
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Palatal Wound
Keywords: Wound Healing; Enamel Matrix Derivative; Palatal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Free Gingival Graft (Sham Comparator): With the aim to ridge preservation after condemned tooth extraction, the socket will be sealed with a free gingival graft removed from the palate. The tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia. After the exodontia, curettage and irrigation of the dental socket will be performed. The free gingival graft will be removed from the donor palatal area with a circular incision of 8 mm and 2 mm thickness. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured. Patient randomized to the Control Group will not receive any kind of treatment in the palatal region.
  Interventions: Procedure: Free gingival graft
- Test Group - Free Gingival Graft + EMD (Experimental): With the aim to ridge preservation after condemned tooth extraction, the socket will be sealed with a free gingival graft removed from the palate. The tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia. After the exodontia, curettage and irrigation of the dental socket will be performed. The free gingival graft will be removed from the donor palatal area with a circular incision of 8 mm and 2 mm thickness. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured. EMD will be applied immediately after the graft removal surgical procedure on the palatal donor area, leaving it in contact with the wound for 5 min. In sequence, it will be covered with an individualized acetate plate that will extend throughout the palatal area and be in position for 2 hours after the procedure
  Interventions: Procedure: Free gingival graft; Device: Enamel Matrix Derivate

INTERVENTIONS:
Procedure: Free gingival graft — Free Gingival Graft removal from the palate donor area for socket preservation
  Other Names: Socket preservation
Device: Enamel Matrix Derivate — EMD in contact with the palate wound for 5 min. After this time, palatal area will be covered with an individualized acetate plate which will stay in position for 2 hours after the procedure
  Arms: Test Group - Free Gingival Graft + EMD

SUMMARY:
The objective of this study is to evaluate clinical and patients-centered parameters of 3-month outcome of the enamel-derived matrix (EMD) application on wound healing process of the donor palatal area after free gingival graft (FGG) removal.

DETAILED DESCRIPTION:
This is a randomized, parallel, double-blind clinical trial. The population that will be evaluated in this is study will be select at Science and Technology Institute - ICT-Sao Jose dos Campos, College of Dentistry.

Patients will be assigned to one of the treatments groups:

* Control Group - Free Gingival Graft (n = 22): Atraumatic extraction surgery and free gingival graft for sealing the entrance of the alveolus
* Test Group - Free Gingival Graft + EMD (n = 22): Atraumatic extraction surgery with placement of a free gingival graft to seal the entrance of the alveolus associated with EMD in the open wound on the palate.

All surgeries will be performed by the same expert periodontist (MMVM). A blade 15c (Swann-Morton® - Sheffield, England) mounted on No. 3 scalpel handle will make an intrasulcular incision around the tooth indicated for exodontia. Then, the tooth will be extracted through the use of appropriate instruments in order to obtain a minimally traumatic exodontia. With the aim to ridge preservation after tooth extraction the socket will be sealed with a free gingival graft removed from the palate. For the free gingival graft removal, a circular template of 8 millimeters in diameter will be used. This stent has the objective of standardizing the palatal graft removal ensuring the wounds will have always the same size. After the circular incision, the graft will be removed with a thickness of 2 millimeters. After free gingival graft removal from palate, it will be adjusted to the entrance of the socket and sutured with Vicryl® 5.0 reabsorbable (Ethicon Johnsons do Brasil, São José dos Campos - SP).

After the graft position, EMD will be applied immediately after the graft removal surgical procedure on the palatal donor area, leaving it in contact with the wound for 5 min. In sequence, it will be covered with an individualized acetate plate that will extend throughout the palatal area and be in position for 2 hours after the procedure.

The evaluated clinical parameters will be: wound remaining area (WRA), scar and tissue colorimetry (TC), tissue thickness (TT) and epithelization (E). Moreover, patient-centered also will be evaluated as: number of pills (NP), tissue edema (TE), postoperative discomfort (D) and Oral Health Impact Profile (OHIP).

All data will be expressed as mean ± standard deviation (SD), and normality will be tested using the Shapiro-Wilk test. Values for remaining wound area, scar and tissue colorimetry, tissue thickness, and epithelization will be examined by repeated measures ANOVA to assess differences within and between groups, followed by a Tukey test for multiple comparisons when the value of p Shapiro-Wilk ≥ 0.05. Those with Shapiro-Wilk p values <0.05 will be analyzed using the Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Values referring to patient-centered parameters such as postoperative discomfort, the number of analgesics taken, tissue edema and oral health impact profile measurements will be analyzed using the T-Test

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 18 years of age, systemically healthy, with good oral hygiene, assessed by plaque index and gingival index of less than 25% (O'Leary et al., 1972);
* Patients with no morphological or pathological changes in the donor palatine region;
* Patients who present an indication of exodontia and with ridge preservation indication for future implantation of implants;
* The tooth included in the study, as well as the adjacent teeth, do not present a loss of periodontal insertion;
* Patients who agreed to and signed the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the present study (Resolution no. 118 - May, 2012, and Ethics and Code of Professional Conduct in Dentistry - 118/12).

Exclusion Criteria:

* Patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers patients;
* Pregnant or lactating patients;
* Patients who had had periodontal surgery on the study area;
* Patients who present opportunistic oral lesions mainly colonized the palate region;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Remaining wound area | 7 days
  The defect area will be measured after 7 post-operative days. For this, standardized photography will be taken ( in terms of brightness, distance and angle). A scale will be used as a reference to measure the area. These photographs will be exported to image software (Image J-NIH, Bethesda, USA) and the wound area will be measured in square millimeters (mm2) (Dias et al. 2015).

SECONDARY OUTCOMES:
Scar and tissue colorimetry | 30 days
  Will be analyzed presence or absence of scar in the operated area after 30 days post-operative. Moreover, Tissue color similarity between the region adjacent to the operated area and the post-operative image were analyzed through photographs. The photographs were exported to image software (Adobe Photoshop 3, München, Germany), and two areas were used: one from the wound and another adjacent area. The areas will be compared ( (ΔE) through the Adobe Photoshop red-green chroma scale and the yellow-blue chroma scale according to the following equation: ΔE =[(L.wound- L.adjacent)2 + (a.wound - a.adjacent)2 + (b.wound - b.adjacent)2] 1/ 2 (Knösel et al., 2009).
Epithelialization | 7 days
  It will be analyzed from the percentage of wound epithelialization (% EF) before the surgical procedure and on 7 days thereafter. The wound will be stained with Shirley's solution (Fig. 8) and the epithelial area will be quantified in the Image J. program. Then, with the total area of the wound, the epithelization% will be calculated (Ozcelik et al. 2008).
Tissue thickness | 90 days
  Tissue thickness of palatine masticatory mucosa will be assessed after 90 days of the procedure. For this, an endodontic spacer with a rubber cursor will be put on the donor area for it to reach the palatine bone plate. Then the cursor will be taken to the tissue, not pressuring it. The distance between the spacer tip and the cursor will be measured using a digital paquimeter (Dias et al. 2015).
Postoperative discomfort | 7 days
  Through air spray for 5 s over the operated site, sensitive function will be measured at 7 days after surgical procedure. After air spray application, patients will be required to use a visual analogue scale (VAS) of 100 mm to assess discomfort; scale extremes will be "no pain" to "extreme."
Number of analgesics | 2 weeks
  Patients will be given a postoperative diary in which they will relate the number of analgesics used during 14 days after the procedure. (Tonetti MS et al. 2017).
Tissue edema | 7 days
  Will be evaluated after 7 days of the surgical procedure with the score: 1 = absent; 2 = slight; 3 = moderate; or 4 = severe (Sanz-Molineret, 2013).
Oral Health Impact Profile | 2 weeks
  Will be evaluated from a questionnaire with 14 questions based on 7 domains: functional limitations, physical pain, psychological discomfort, physical disability, psychological deficiency and social deficiency. The patient should respond to the questions within 14 days after the surgical procedure, performing a postoperative diary. For each question an answer must be given, represented in numbers, being: 0- Never; 1- Almost never; 2-Occasionally; 3-Quite frequent; 4-Very common; 5-I do not know (Tonetti MS et al. 2017).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT- UNESP
Locations (1):
- Manuela Maria Viana Miguel, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nokhbehsaim M, Winter J, Rath B, Jager A, Jepsen S, Deschner J. Effects of enamel matrix derivative on periodontal wound healing in an inflammatory environment in vitro. J Clin Periodontol. 2011 May;38(5):479-90. doi: 10.1111/j.1600-051X.2010.01696.x. Epub 2011 Jan 16. PMID 21235616
- [Background] Miron RJ, Dard M, Weinreb M. Enamel matrix derivative, inflammation and soft tissue wound healing. J Periodontal Res. 2015 Oct;50(5):555-69. doi: 10.1111/jre.12245. Epub 2014 Nov 23. PMID 25418917